CLINICAL TRIAL: NCT01044485
Title: A Multicenter Open-label, Phase I/II Dose Escalation Study of Oral Lapatinib in Combination With Docetaxel in Patients With HER-2 Positive Advanced or Metastatic Breast Cancer
Brief Title: Lapatinib in Combination With Docetaxel in Patients With HER-2 Positive Advanced or Metastatic Breast Cancer
Acronym: LapDoc
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Collaborators: GlaxoSmithKline (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0205-1isni 07 / 001.112
Record Dates: First submitted 2010-01-05; First posted 2010-01-08 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Metastatic Breast Cancer
Keywords: HER-2 positive advanced or metastatic breast cancer; dose escalation study; lapatinib; docetaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lapatinib + docetaxel (Other): dose level Lapatinib (OD) Docetaxel (q3wks) Systematic Growth factor Minus 0 1250 mg 75 mg/m2 + systematic growth factor support
  0, 1250mg 75 mg/m2 No
  +1 1500mg 75mg/m2 No
  Minus +1* 1500mg 75mg/m2 + systematic growth factor support
  +2 1250mg 100mg/m2 No
  Minus +2* + systematic growth factor support
  +3 1500mg 100mg/m2 No
  Minus +3* + systematic growth factor support
  Apart within the minus dose levels, G-CSF support should be added only as rescue strategy if severe neutropenia occurred during the first cycle of studied dose.Patients will receive 4 cycles of the association. In case of benefit of the treatment, they should continue the treatment with lapatinib until progression.* patients will be included at level "minus X" only if 2 DLT out of 6 patients based on febrile neutropenia occurred at level "X"
  Interventions: Drug: lapatinib; Drug: docetaxel

INTERVENTIONS:
Drug: lapatinib — escalation dose from 1250 to 1500 mg in association with docetaxel
Drug: docetaxel — escalation dose from 75 mg/m2 to 100 mg/m2 in association with lapatinib

SUMMARY:
The objective of this phase I/ II study is therefore to assess the safety and efficacy of lapatinib in combination with docetaxel in patients with advanced cancer. Only patients in first line treatment for metastatic disease should be included in the present study. It is proposed to start with a phase I part evaluating the safety of lapatinib 1250 mg with docetaxel 75 mg/m² without systematic support of growth factors, starting after the completion and data from the 1000 mg lapatinib +75 mg/m² docetaxel dose level in the EORTC (Bonnefoi) study.The objective of the phase II part will confirm the safety and evaluate efficacy of lapatinib in combination with docetaxel.

DETAILED DESCRIPTION:
Docetaxel is a major drug in the treatment of metastatic breast cancer. In HER2 negative tumor, the first line treatment is based on docetaxel containing regimen: docetaxel alone, docetaxel + anthracycline or docetaxel + capecitabine. The efficacy of docetaxel in combination with trastuzumab has been demonstrated in first line metastatic breast cancer overexpressing erbB2 receptor. The response rate (RR) and the time to progression (TTP) observed were even higher than those obtained with paclitaxel +trastuzumab. Docetaxel is more and more used in first line metastatic setting, becoming the first Taxane used in this setting.As trastuzumab may raise safety/tolerability concerns, and as its interest in trastuzumab refractory patients may be limited, there is a need to find new drugs to combine with docetaxel in breast cancer, and to address the specific interaction/safety profile of this combination.The association of lapatinib and docetaxel will be the key combination in metastatic breast cancer development for GSK.The conclusion of a phase I trial EGF 10021 trial conducted in the US which assessed the combination of lapatinib and docetaxel showed that the acceptable optimal tolerated regimen (OTR) of docetaxel (75 mg/m²) was obtained in combination with lapatinib 1250 mg with systematic growth factor support.Data from an ongoing EGF100161 phase I study evaluating the OTR of lapatinib + docetaxel + trastuzumab shows that the association of lapatinib 1250 mg with docetaxel 75mg/m² is haematological toxic and has recently been amended to evaluate lapatinib 1250 mg with docetaxel 75 mg/m² with systematic growth factor support.A phase I/II EORTC study evaluating docetaxel plus lapatinib in neoadjuvant breast cancer patients has just started. The phase I part of this study will evaluate several lapatinib and docetaxel dose levels before conducting phase II.

The phase I part will enrol patients (in cohorts of 3 or 6) to determine in a step-wise approach, the OTR of lapatinib and docetaxel. Patients should not be entered at a higher dose level until all patients in the previous cohort complete the first cycle of treatment, this first cycle is used to determine OTR. Dose modification of lapatinib will be based on any observed toxicity in the treatment period. The OTR will be defined as the dose level at which £ 1 of 6 patients experiences the DLT (dose limiting toxicity).If no DLT is observed in the first 3 patients at a particular dose level during the first cycle (3 week treatment period), recruitment will start at the next dose levelIf 1/3 patients experiences a DLT at a particular dose level, additional 3 patients will be enrolled at that dose level to a total of 6 patients if no DLT occurred againIf 1/6 patients experiences a DLT at a particular dose level, recruitment will start at the next dose levelIf ³ 2/6 patients experiences the same DLT at a particular dose level, the dose level is not considered to be tolerableIf ³ 2/6 patients experiences two distinct DLT at a particular dose level, additional 3 patients will be enrolled at that dose level to a total of 9 patients. If one of the previously described DLT occurred again among the new enrolled patients, the dose level is not considered to be tolerableA total of 12 patients will be treated at the OTR.The OTR is defined as the dose level at which no more than 1 of 6 patients experiences a DLT.The DLT for this study is defined during cycle 1 for the dose escalation step as:· any grade 3-4 non hematological toxicity as defined by the Common Toxicity Criteria, version 3 (with the exclusion of alopecia, nausea, vomiting, diarrhea, infusion related that can be rapidly controlled with appropriate measures)· an absolute neutrophil count (ANC) < 0.5x109 /L lasting for > = 7 day· febrile neutropenia defined as ANC < 1.0 x109 /L and fever at least 38.5°C· thrombocytopenia < 25, 000/µl or thrombocytopenic bleeding requiring transfusion· grade 3 or higher left ventricular cardiac dysfunction or a ≥ 20% decrease from baseline in left ventricular ejection fraction (LVEF) that is also below the institution's lower limit of normal (LLN), and confirmed by a repeat evaluation 1 to 2 weeks following the first evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age over or equal 18 years·
* ECOG Performance Status of 0 to 2·
* Patients with histological or cytological confirmed breast cancer, HER positive (IHC 3+, or IHC 2+ and FISH/CISH +, or FISH+ or CISH+ only), not amenable for an alternative curative strategy in first line metastatic setting·
* Patients who receive hormonotherapy for metastatic disease or who received chemotherapy in adjuvant setting if recurrence occur after 6 months are eligible·
* Patient must have not received the last injection of trastuzumab within the six weeks·
* Subjects must have completed prior radiotherapy treatment at least 4 weeks from enrolment and recovered from all treatment-related toxicities· Subjects must have tissue available to prospectively determine treatment assignment and to compare tumor response with intra-tumor expression levels of relevant biomarkers·
* No prior systemic investigational agent within the past 30 days or topical investigational drugs within the past 7 days·
* Subjects must have a cardiac ejection fraction within the institutional range of normal as measured by ECHO (echocardiogram) or MUGA (Multigated Acquisition) scan·
* Subjects must have adequate haematological, hepatic, and renal function·
* Affiliation to a social insurance program is required

Exclusion Criteria:

* Subjects with elevations of transaminase (ALT and/or AST) greater than 2.5 times the upper limit of the normal range (ULN) are NOT eligible for the study·
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier·
* Patients who have had prior treatment with EGFR targeting therapies· All herbal (alternative) medicines are excluded·
* Patients with known brain metastases·
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib.·
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, peripheral neuropathy of grade 2 or greater, or psychiatric illness/social situations that would limit compliance with study requirements·
* Pregnant women are excluded from this study because lapatinib is member of the 4-anilinoquinazoline class of kinase inhibitors with the potential for teratogenic or abortifacient effects·
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with lapatinib·
* Patients with gastro intestinal (GI) tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)· Current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)· Previous allergic reaction to docetaxel and/or polyascorbate· Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors·
* Active cardiac disease, defined as: history of uncontrolled or symptomatic angina pectoris, history of cardiac arrhythmias requiring medications, or clinically significant, with the exception of asymptomatic atrial fibrillation requiring anticoagulation, myocardial infarction < 6 months from study entry, uncontrolled or symptomatic congestive heart failure, ejection fraction below the institutional normal limit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-11; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To determine the optimal tolerated regimen of lapatinib administered in combination with docetaxel as first-line therapy in patients with metastatic breast cancer | during first cycle ( each cycle last 3 weeks)

SECONDARY OUTCOMES:
To evaluate the dose-limiting toxicity | each weeks of each cycle and after the end of the study
To evaluate anti-tumour activity in terms of response | each cycle and at the end of the study
To evaluate anti-tumour activity in time to response | each cycle and at the end of the study
To evaluate anti-tumour activity in terms of response duration | each cycle and at the end of the study
To evaluate anti-tumour activity, in terms time to progression (TTP) | each cycle and at the end of the study
To evaluate anti-tumour activity, in terms of time to treatment failure (TTF) | each cycle and at the end of the study
To evaluate anti-tumour activity, in terms of overall survival (OS) | at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Isambert, MD, Principal Investigator — Centre Georges François Leclerc
Locations (1):
- Centre Georges François Leclerc, Dijon, Bourgogne-Franche-Comté, France